CLINICAL TRIAL: NCT05901207
Title: Diagnostic and Prognostic Biomarkers for IgG4-related Disease.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-EIG-2022-92
Record Dates: First submitted 2023-01-11; First posted 2023-06-13 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2023-06

CONDITIONS: Immunoglobulin G4-Related Disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case
  Interventions: Diagnostic Test: blood test

INTERVENTIONS:
Diagnostic Test: blood test — blood test

SUMMARY:
IgG4-immunoglobulin-related disease (IgG4-IRD) is a relatively new pathology, characterized by intense inflammation, fibrosis, infiltration and elevated IgG4 levels in peripheral blood.

Despite the interest in the disease, these diagnostic criteria are not without discrepancies and false negatives. In fact, despite the fact that elevated serum IgG4 concentrations can provide an important clue for the diagnosis of the disease,described that the specificity and positive predictive value of elevated serum IgG4 concentrations are 60 % and 34 % respectively. And, when they increased the cut-off values to double to improve specificity, the sensitivity of IgG4 levels drops to 35 %.

In 2014, was described the presence of elevated concentrations of plasmablasts (CD19 low, CD20 -, CD38+ and CD27+) in the serum of patients with active ER-IgG4, even in patients with normal IgG4 levels, compared with healthy patients and with other autoimmune pathologies.

Furthermore, several studies have shown that follicular T helper (Thf) cells are increased in both peripheral blood and affected tissue of patients with ER-IgG4. These cells appear responsible for the development of germinal centers in lymph nodes and for the production of interleukins that drive IgG4 class switching, and creation of IgG4-secreting plasmablasts and plasma cells. This suggests that interleukins IL4, IL5, IL 10, IL13 might also be relevant in discerning ER-IgG4 from other immune-mediated processes with similar symptoms.

ACTION GOALS:

1. To evaluate the diagnostic validity of plasmablast count and other immunological markers (B lymphocyte differentiation stage, follicular T helper lymphocytes (Thf) and IL-4, IL5, IL-10 and IL-13) in peripheral blood for IgG4-Related Disease.
2. To evaluate the correlation of these biomarkers with inflammatory activity, clinical manifestation and diagnostic certainty (possible, probable or definite) of IgG4-Related Disease.
3. To evaluate whether high counts or concentrations of these biomarkers at diagnosis are prognostic factors for relapse during the first 12 months of follow-up in patients with IgG4-Related Disease.

DETAILED DESCRIPTION:
1. Project design The project will consist of a first diagnostic study (objectives 1-2) of cross-sectional analytical design to assess the validity of the biomarkers. Subsequently, a second prospective cohort study (objective 3) will be carried out to evaluate whether these biomarkers are prognostic factors for relapse in patients with IgG4-related disease after treatment.
2. Scope of the project The project will be carried out at the Hospital Sant Pau which is a tertiary referral center of the AIS Dreta (Área Integral de Salud) of Barcelona. The hospital covers a population of 407,550 inhabitants. IgG4-Related Disease is a rare disease that requires diagnostic tests and treatments for hospital use, so almost all cases are referred and followed up at the hospital. At the Functional Autoimmune Unit of the Hospital de Sant Pau the investigators perform monographic consultations on systemic vasculitis, the investigators are an active part of the Aortic Pathology Unit (source of patients with aortitis and retroperitoneal fibrosis), and the investigators maintain a close relationship with the other services involved in this pathology (otorhinolaryngology, digestive and nephrology).
3. Period of performance and recruitment procedure Patients will be selected by sequential sampling between April 2023 and December 2023 in the Systemic Autoimmune Diseases monographic consultations.
4. Sample size IgG4-related disease is a rare disease and has therefore been defined under a pragmatic and realistic approach. A total of 50 participants will be recruited at Hospital Sant Pau in Barcelona. It is planned to recruit 50 patients with IgG4 disease which would be the totality of newly diagnosed patients during 12 months in our center and 50 patients with osteoarthritis or soft tissue pathology. In a previous study (doi: 10.1097/MD.00000000000000003785) the correlation of serum IgG4 concentration with active disease was r=0.17 while the correlation of IgG4+ plasmablasts (10.1136/annrheumdis-2014-205233) with active disease was r=0.47. The expected size to detect a difference (r1-r) of 0.28 is 84 patients with a beta of 20% and alpha of 5%.
5. Data collection Data will be collected from the electronic medical record of the hospital database.

   * Demographic and disease assessment: Collection of demographic (age, sex) and disease information (onset, duration of symptoms, treatments). Disease onset will be defined as the time at which ER- IGg4 diagnostic counseling is performed according to the Umehara criteria. The status of the outcome event (disease relapse) and the date on which it occurs will be collected. The start date of follow-up, date of outcome event, last follow-up visit or last contact with the patient in the case of lost subjects will be collected.
   * Clinical evaluation: The clinical evaluation will be carried out according to medical criteria, taking into account the combination of the patient's clinical status and the complementary radiological and serological examinations, classifying the patient as active or inactive.
   * Radiological studies: Data from radiological examinations in the form of CT and/or FDG18F-PET/CT performed in the diagnosis and/or evolutionary control of the patients will be collected. The organs affected and the increase of 18F FDG in case of PET-CT will be taken into account. In those patients who have scans at diagnosis and control visits, a qualitative comparative study of the images will be performed (no change, improvement, worsening).
   * Laboratory studies: Plasmablasts are one of the differentiation stages of B lymphocytes. At the peripheral blood level, the investigators can identify them by labeling against molecules on their surface. Plasmablasts are defined as CD45+ CD19+ IgM- IgD- CD27+ CD38high cells. The use of these markers also allows us to identify other differentiation stages such as naïve B lymphocytes (CD45+ CD19+ IgD+ CD27-), marginal zone (CD45+ CD19+ IgD+ CD27+), class non-switched (CD45+ CD19+ IgM+ IgD+ IgD+ CD27+ CD38-), class switched memory (CD45+ CD19+ IgM- IgD- CD27+ CD38-), transitional (CD45+ CD19+ IgM+ IgD+ CD27- CD38high CD24high), CD19low (CD45+ CD19low CD27+) or CD21low (CD45+ CD19+ CD21low CD38-).

   To analyze the differentiation stages of B lymphocytes, the investigators will perform a flow cytometry analysis. Briefly, from peripheral blood in EDTA, the investigators will perform a wash and subsequent staining with the different monoclonal antibodies directed against the surface molecules of interest labeled with fluorochromes. After a 15-minute incubation, the red blood cells are lysed, washed again and analyzed in the BD FACSLyric cytometer.

   For the determination of follicular T helper (Thf) lymphocytes and Thf1 and Thf2 subpopulations the investigators will also perform cytometry analysis with monoclonal antibody staining, defining Tfh1 as CD4+ CD45RA- CXCR5+ CCR6- CXCR3+ T lymphocytes and Tfh2 as CD4+ CD45RA- CXCR5+ CCR6- CXCR3- T lymphocytes.

   The analysis of interleukins IL-4, IL-5, IL-10 and IL-13 will be performed, from our serum, by individualized ELISAs for each of them.

   The analysis of the biosamples and images will be performed at the research center (Hospital Sant Pau de Barcelona).
6. Description of variables 6.1. Baseline study

   * Dependent or response variables: Disease activity, prevalence of IgG4-related disease according to different degrees of diagnostic certainty, type of clinical manifestation, number of organs affected, IGg4 concentration and acute phase reactants.
   * Independent variables: plasmablast count, differentiation stages of B lymphocytes and Thf lymphocytes in peripheral blood and serum concentration of interleukins (IL-4, IL-5, IL-10 and IL-13).

   6.2. Longitudinal study
   * Response-dependent variables: Disease relapse and persistence of disease activity will be studied according to medical criteria.
   * Independent variables: plasmablast count, differentiation stages of B lymphocytes and Thf lymphocytes in peripheral blood and serum concentration of interleukins (IL-4, IL-5, IL-10 and IL-13).
   * Potentially confounding variables: Demographics (age, sex, race), IgG4-related disease subtype according to organ specificity, number of organs affected, time from onset of symptoms and time to initiation of treatment, accumulated corticosteroid dose, immunomodulatory or biological treatment.
7. Follow-up At the baseline visit, demographic and disease information will be collected in a standardized manner. Blood sampling is performed within 30 days as per standard clinical practice. Imaging tests such as CT or PET-CT are usually performed 1 month before or after the baseline visit. Follow-up visits will be performed every 4 months per usual clinical practice without requiring additional visits except for those presenting complications or adverse effects to the treatments.
8. Statistical analysis Logarithmic transformation of biomarker levels will be performed if they do not follow a normal distribution.

   * Objectives 1 and 2: Sensitivity, specificity and area under ROC curve will be calculated. Pearson's or Spearman's correlation coefficient will be used according to applicability conditions.
   * Objective 3: Univariate Cox regression will be performed to evaluate the prognostic value of biomarkers for predicting relapse. Survival will be defined as the time between the baseline visit at diagnosis to the date of the outcome event (relapse or persistence of inflammatory activity). Median follow-up will be calculated according to the inverse Kaplan Meier method. Other factors that may be related to survival (biological treatment, cumulative corticosteroid dose, age, acute phase reactants) will be added. Binary logistic analysis will also be performed to assess the association between biomarkers and dependent variables. The significance level will be set at 5% bilaterally. The statistical program Stata 14.0 for Windows will be used.
9. Ethics The study will be conducted in strict accordance with international ethical recommendations for medical research in humans. The investigator will be responsible for ensuring that the study is conducted in accordance with the Bioethical Research Law 14/2007. Before starting the study, the Ethics Committee of the investigating Hospital must approve the study protocol, the information to be given to the subject and the informed consent form to be used. The CEIC will be informed of any subsequent amendments to the protocol and must be asked for its opinion in the event that a new evaluation of the ethical aspects of the study is necessary. Regarding the confidentiality of the study data, the provisions of the Organic Law 3/2018 of December 5, "Protection of Personal Data" will be followed. Your name will not appear in any of the study reports and your identity will not be disclosed to any person except to fulfill the purposes of the study, and in the case of medical emergency or legal requirement.
10. Limitations Because it is a rare disease, the sample size is the main limitation of the study and will limit the number of variables that can be included in the analysis. In order to address this limitation, the investigators will disseminate the present study in the rest of the services and multidisciplinary meetings of our center, making an active search for possible candidates to be included in the study. Another limitation is that the diagnosis of the cases is defined by clinical criteria, not always confirmed histopathologically. This is an unavoidable limitation due to the clinical nature of the study. For this reason it was decided to opt for a prospective design compared to many studies of histopathologically confirmed cases that are usually retrospective. Finally, the results will not be validated in an independent sample so the results must be interpreted in context.
11. CHRONOGRAM The total duration of the project is 2 years; 18 months for field work with recruitment and inclusion of patients and processing of biological samples. The last 6 months are reserved for the analysis, interpretation and writing up of results.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Diagnosed of IgG4-related disease (possible, probable or definite) according to the revised Umehara diagnostic criteria

Exclusion Criteria:

* Patients with cancer
* secondary causes of fibrosis
* Granulomatosis
* Castleman's disease
* seropositive Sjögren's syndrome
* Primary sclerosing cholangitis.
* Patients who have received treatment with prednisone ≥ 5 mg, immunosuppressive or biologic treatment in the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the monographic consultations of systemic autoimmune disease of a tertiary university, Hospital Universitari Sant Pau
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-02 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in IgG4 in peripheral blood | Change from Baseline at one year after the study began
  g/L Independent variables: plasmablast count, differentiation stages of B lymphocytes and Thf lymphocytes in peripheral blood and serum concentration of interleukins (IL-4, IL-5, IL-10 and IL-13).
  and serum concentration of interleukins (IL-4, IL-5, IL-10 and IL-13).
Change in IL-4 | Change from Baseline at one year after the study began
  pg/mL
Change in IL-5 | Change from Baseline at one year after the study began
  pg/mL
Change in IL-10 | Change from Baseline at one year after the study began
  pg/mL
Change in IL-13 | Change from Baseline at one year after the study began
  pg/mL
Change in plasmablast | Change from Baseline at one year after the study began
  SFU/million

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Moya Alvarado, Principal Investigator — Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Carruthers, M. N., Khosroshahi, A., Augustin, T., Deshpande, V., & Stone, J. H. (2015). The diagnostic utility of serum IgG4 concentrations in IgG4-related disease. Annals of the Rheumatic Diseases, 74(1), 14-18. — https://doi.org/10.1136/annrheumdis-2013-204907
- See also: Hong, X., Li, W., Xie, X.-Y., Zhang, Z.-Y., Chen, Y., Gao, Y., Peng, X., Su, J.-Z., Zhang, Y.-Y., Wang, Z., Cai, Z.-G., Zhang, L., Liu, Y.-Y., He, J., Ren, L.-M., Li, Z.-G., & Yu, G.-Y. (2017). Differential diagnosis of IgG4-related sialadenitis, primary — https://doi.org/10.1016/j.bjoms.2016.10.021
- See also: Maehara, T., Pillai, S., Stone, J. H., & Nakamura, S. (2019). Clinical features and mechanistic insights regarding IgG4-related dacryoadenitis and sialoadenitis: a review. International Journal of Oral and Maxillofacial Surgery, 48(7), 908-916. — https://doi.org/10.1016/J.IJOM.2019.01.006
- See also: Okazaki, K., Uchida, K., Koyabu, M., Miyoshi, H., & Takaoka, M. (2011). Recent advances in the concept and diagnosis of autoimmune pancreatitis and IgG4-related disease. Journal of Gastroenterology, 46(3), 277-288. — https://doi.org/10.1007/s00535-011-0386-x